CLINICAL TRIAL: NCT02826980
Title: Observational Study Rheumatological Manifestations Associated With Endometriosis
Acronym: ENDOMETRIOS
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOMETRIOS
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatology; Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire — Patients consultant in gynecology in the service of Doctor Sauvanet, for whom a diagnosis of endometriosis has been established (clinical history and imaging tests confirming the diagnosis) will be offered to fill a self-administered questionnaire during their consultation

SUMMARY:
Endometriosis is defined as the presence of endometriotic tissue outside the uterus. Its pathophysiology is still misunderstood today, but more and more work on this pathology are published. The clinical presentation is generally characterized by the existence of cyclical pelvic pain, with dysmenorrhea, dyspareunia, dysuria, dyschezia.

But, there are a wide variety of symptoms, with different painful sites and different types of pain.

The estimated prevalence of endometriosis is about 10% in women. But the impact of this disease on quality of life and its economic impact is estimated considerable. In a US study, the direct costs associated with endometriosis were estimated at US $ 2.801 per woman. Some studies have focused also to quantify work absenteeism associated with endometriosis.

The etiology of endometriosis is based on the migration of endometrial fragments reaching the pelvis via the tubes and establishing themselves on other sites, thus creating non cyclical uterine pain. Catamenial pace of pain is suggestive of the diagnosis, but with time, the pain tends to be chronic rather than cyclical. The standard diagnosis is based on visualization and histological examination of the lesions.

The wide variety of symptoms of endometriosis often leads to wandering and medical diagnostic delay. A better understanding of this disease by the medical community would allow better management of these patients. Currently, endometriosis remains a misunderstood disease by rheumatologists. However, the initial presentation may mimic rheumatologic symptoms; thus, rheumatologists may face this disease.

The purpose of this study was to determine the prevalence and characteristics of manifestations of endometriosis in a cohort of patients with a recent diagnosis of endometriosis established. Secondly, it may well be possible to establish a list of symptoms and signs suggestive of endometriosis for the rheumatologist, allowing to contact a specialized consultant gynecologist some patients "by mistake" in rheumatology.

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometriotic tissue outside the uterus. Its pathophysiology is still misunderstood today, but more and more work on this pathology are published. The clinical presentation is generally characterized by the existence of cyclical pelvic pain, with dysmenorrhea, dyspareunia, dysuria, dyschezia.

But, there are a wide variety of symptoms, with different painful sites and different types of pain.

The estimated prevalence of endometriosis is about 10% in women. But the impact of this disease on quality of life and its economic impact is estimated considerable. In a US study, the direct costs associated with endometriosis were estimated at US $ 2.801 per woman. Some studies have focused also to quantify work absenteeism associated with endometriosis.

The etiology of endometriosis is based on the migration of endometrial fragments reaching the pelvis via the tubes and establishing themselves on other sites, thus creating non cyclical uterine pain. Catamenial pace of pain is suggestive of the diagnosis, but with time, the pain tends to be chronic rather than cyclical. The standard diagnosis is based on visualization and histological examination of the lesions.

The wide variety of symptoms of endometriosis often leads to wandering and medical diagnostic delay. A better understanding of this disease by the medical community would allow better management of these patients. Currently, endometriosis remains a misunderstood disease by rheumatologists. However, the initial presentation may mimic rheumatologic symptoms; thus, rheumatologists may face this disease.

The purpose of this study was to determine the prevalence and characteristics of manifestations of endometriosis in a cohort of patients with a recent diagnosis of endometriosis established. Secondly, it may well be possible to establish a list of symptoms and signs suggestive of endometriosis for the rheumatologist, allowing to contact a specialized consultant gynecologist some patients "by mistake" in rheumatology.

Main objective / secondary:

Observational study rheumatological manifestations associated with endometriosis: prevalence and characteristics of rheumatological manifestations associated with endometriosis, via a self-administered questionnaire.

Methodology :

Design: Prospective, observational Time study: 3 to 6 months

Acquisition of data:

* Self-administered questionnaire (in PJ)
* Supports state and annex: FIU PJ, Excel grid of data collection.
* Statistical analysis Saint Joseph
* Clarify data anonymisation: not anonymisation, but confidentiality.

Development of the study:

- Describe how the study:

Patients consultant in gynecology in the service of Doctor Sauvanet, for whom a diagnosis of endometriosis has been established (clinical history and imaging tests confirming the diagnosis) will be offered to meet a self-administered questionnaire during their consultation. This will be delivered by the gynecologist in the consultation, with the consent sheet. If the patient agrees, the self-administered questionnaire must be completed in the consultation box or in the waiting room, and handed to the gynecologist or the secretary of the consultation.

Data will be collected and analyzed.

- Expected duration of patient recruitment: 3 months

ELIGIBILITY:
Inclusion Criteria:

* Women with endometriosis diagnosis established and confirmed at St. Joseph Hospital.

Exclusion Criteria:

* aged <18 yo and menopause or aged >50 yo

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with endometriosis diagnosis established and confirmed consulting at St. Joseph Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Endometriosis stage | Day 1
  According to the classification of the AFS (American Fertility Society)

SECONDARY OUTCOMES:
Rheumatic stage | Day 1
  Radiographic stages of knee OA:
  0 normal radiographic stage Stage 1 of questionable significance osteophytes Stage 2 net osteophytes without changing the joint line Stage 3 net decrease osteophytes and joint space Stage 4 Severe narrowing of the joint space and sclerosis of the subchondral bone.
  Radiological stages of osteoarthritis:
  Stage 0 normal radiographic Stage 1 joint space narrowing, osteophytes doubtful péricapitale Stage 2 joint space narrowing, osteophytes, moderate bone sclerosis Stage 3 net joint space with discrete osteophytes, bone sclerosis with cyst deformation of the femoral head and acetabulum minimal Stage 4 dispariton joint space with bone sclerosis and cyst, significant deformation of the femoral head and the acetabulum, with major osteophytes.
Analogic Pain Evaluation | Day 1
  On a scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: PORTIER Agnes, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France